CLINICAL TRIAL: NCT05353374
Title: Effectiveness of Sodium Fusidate Ointment Compared to Petrolatum for Wound Healing Following Cauterization: A Double-Blind Randomized Controlled Trial
Brief Title: Effectiveness of Sodium Fusidate Ointment Compared to Petrolatum for Wound Healing Following Cauterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Firman Parrol, Dermatology Resident, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-11-1406
Record Dates: First submitted 2022-04-23; First posted 2022-04-29 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Seborrheic Keratosis; Acrochordon
Keywords: wound healing; cauterization; sodium fusidate ointment; petrolatum
MeSH Terms: conditions — Keratosis, Seborrheic | interventions — Fusidic Acid; Ointments

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Allocation sequence was generated by a statistician with a computer and it was concealed from the researchers and participants. The ointment was prepared and packaged by a pharmacist. Each pot was numbered in accordance with the allocation sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium fusidate ointment (Experimental): Electrosurgery was carried out using Ellman® Surgitron. The tissue was cleaned using sterile gauze or a cotton swab that had been moistened with 0.9% NaCl. Following electrosurgery, sodium fusidate ointment was applied to the wound according to the allocation sequence. The patient also received a wound care instruction sheet. Each subject was given two or four pots of ointment that should be applied twice daily on the wound.
  Interventions: Drug: Sodium Fusidate 2 % Topical Ointment
- Petrolatum (Placebo Comparator): Electrosurgery was carried out using Ellman® Surgitron. The tissue was cleaned using sterile gauze or a cotton swab that had been moistened with 0.9% NaCl. Following electrosurgery, petrolatum was applied to the wound according to the allocation sequence. The patient also received a wound care instruction sheet. Each subject was given two or four pots of ointment that should be applied twice daily on the wound.
  Interventions: Drug: Petrolatum ointment

INTERVENTIONS:
Drug: Sodium Fusidate 2 % Topical Ointment — Sodium fusidate 2% topical ointment was applied twice daily on the wound after cauterization for 14 days.
  Other Names: Fucidin ointment
  Arms: Sodium fusidate ointment
Drug: Petrolatum ointment — Petrolatum ointment was applied twice daily on the wound after cauterization for 14 days.
  Other Names: Vaseline album
  Arms: Petrolatum

SUMMARY:
A double-blind within person randomized controlled trial study was conducted on 90 wounds in 22 subjects. All wounds were randomized to receive either sodium fusidate ointment or petrolatum following cauterization.

DETAILED DESCRIPTION:
All eligible participants were randomized to be applied sodium fusidate ointment (intervention) or white petrolatum (control) on the lesions on their face with 1:1 ratio. Allocation sequence was generated by a statistician with a computer and it was concealed from the researchers and participants. The ointment was prepared and packaged by a pharmacist. Each pot was numbered in accordance with the allocation sequence.

Electrosurgery was carried out using Ellman® Surgitron. Prior to the cauterization, we performed infiltration anesthesia around the lesion with Pehacain® (containing 20 mg of lidocaine and 0.0125 mg/ml epinephrine). The tissue was cleaned using sterile gauze or a cotton swab that had been moistened with 0.9% NaCl. Following electrosurgery, sodium fusidate ointment or petrolatum was applied to the wound according to the allocation sequence. The patient also received a wound care instruction sheet. This sheet contained information on how to wash the face or body properly, how to apply the ointment properly, what to avoid after procedure (rubbing the wound excessively, use make up, sweating excessively, and use other topical agents on the wound), and follow-up instructions (on the 3rd, 7th, and 14th day). Each subject was given two or four pots of ointment that should be applied twice daily on the wound.

Wound monitoring, which includes erythema, edema, crusting, re-epithelialization, total wound healing score, pus, and subjective symptoms was performed on the 3rd, 7th, and 14th day. Erythema scores was also monitored immediately after electrosurgery. Monitoring can be done 1 day earlier or later than schedule in some cases since the wound healing phase is expected still the same. Clinical grading of each site was carried out using a 5-point analog scale for erythema, edema, crusting, re-epithelialization, and total wound healing score.

ELIGIBILITY:
Inclusion Criteria:

* age over 20 years
* clinically diagnosed with seborrheic keratosis or acrochordon
* having minimum of two lesions and maximum of four lesions with diameter of 4-10 mm on face or neck and minimum distance between lesions of 5 cm
* providing consent to participate into the study

Exclusion Criteria:

* a skin bacterial infection on the other parts of body's skin
* benign tumor lesions with inflammation or secondary infection
* history of antibiotics use in the last 2 weeks or long-acting penicillin injections within the past 1 month
* history of corticosteroids and immunosuppressants use in the past 2 weeks
* using a pacemaker
* infected with Coronavirus disease 2019 (Covid-19).

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Wound healing score | 14 days
  Wound healing score was calculated based on the erythema, edema, crusts, and reepithelization. Wound healing score is as follows: 0-4 = very good/healed, 5-8 good/healed, 9-12 moderate/not healed, and 13-16 = poor/not healed

SECONDARY OUTCOMES:
Erythema | 14 days
  Skin erythema around the wound, assessed with physical examination. Erythema score is as follows: 0 = no erythema, 1 = mild erythema (25%), 2 = moderate erythema (50%), 3 = severe erythema (75%), and 4 = very severe erythema (100%)
Edema | 14 days
  Edema on the wound area, assessed with physical examination. Edema score is as follows: 0 = no edema, 1 = mild edema (25%), 2 = moderate edema (50%), 3 = severe edema (75%), and 4 = very severe edema (100%)
Crusts | 14 days
  Presence of crusts on the surface of the wound, assessed with physical examination. Crusts score is as follows: 0 = none, 1 = a few (1-30%), 2 = moderate (31-60%), 3 = a lot (61-90%), and 4 = generalized (91-100%)
Reepithelization | 14 days
  Improvement of the wound characterized by decreasing size and depth of the wound, assessed with physical examination. Reepithelization score is as follows: 0 = complete (91-100%), 1 = good (61-90%), 2 = moderate (1-30%), and 4 = poor (0% or widening of the wound)
Incidence of infection | 14 days
  Presence of wound infection, established by findings of pain, erythema, edema, and poor reepithelization

CONTACTS AND LOCATIONS:
Overall Officials: Firman Parrol, MD, Principal Investigator — Indonesia University
Locations (1):
- Dermatology and Venereology Clinic, Dr. Cipto Mangunkusumo National Central General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No